CLINICAL TRIAL: NCT03593837
Title: A Multicenter, Randomized, Double-blind,Placebo-controlled Trial Evaluating the Efficacy and Safety of Huang Qi GuiZhi Wu Wu Tang Granulesin Patients With Rheumatoid Arthritis
Brief Title: Efficacy and Safety of HQGZWWT Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cui xuejun (Other)
Responsible Party: Sponsor-Investigator, Cui xuejun, Principal Investigator base of Traditional Chinese Medicine, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HQGZWWT
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Huang Qi Gui Zhi Wu Wu Granule; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients are given HQGZWWT granules (orally twice a day for 3 months and instructed to dissolve one package (4 g) with hot water (200 mg).
  Interventions: Drug: Huang qi gui zhi wu wu granule
- Placebo group (Placebo Comparator): Patients are given HQGZWWT granules placebo (orally twice a day for 3 months and instructed to dissolve one package (4 g) with hot water (200 mg).
  Interventions: Drug: Huang qi gui zhi wu wu granule placebo

INTERVENTIONS:
Drug: Huang qi gui zhi wu wu granule — Patients are given HQGZWWT granules (orally twice a day for 3 months and instructed to dissolve one package (4 g) with hot water (200 mg)
  Arms: Experimental group
Drug: Huang qi gui zhi wu wu granule placebo — Patients are given HQGZWWT granules placebo (orally twice a day for 3 months and instructed to dissolve one package (4 g) with hot water (200 mg)
  Arms: Placebo group

SUMMARY:
Rheumatoid arthritis (RA) is a chronic autoimmune disease characterized by swelling, pain, and synovial damage. Effective methods lack in the treatment of RA. A traditional prescription in use for thousands of years in China, Huang Qi Gui Zhi Wu Wu Tang(HQGZWWT)granule is still chosen to relive pain and prevent joint malformation in RA patients. However, no evidence-based medical research has been organized to assess the effectiveness and safety of HQGZWWT granules for RA.

DETAILED DESCRIPTION:
Investigators will conduct a multicenter, randomized, double-blind, placebo-controlled clinical trial to determine whether HQGZWWT granules can relieve pain and protect joints. Investigators will randomly divide 120 patients with active arthritis for 3 months. Main measurements include ratio of 50 of ACR (American College of Rheumatology), change of DAS (28) from baseline to 3 months, and SHARP scores of van der Heijde from baseline to 12 months. SecondarymeasurementsincludeACR20, ACR70, Health Assessment Questionnaire-Disability Index (HAQ-DI), arthritis pain score, and Patient Global Assessment of Arthritis. The time points are set as baseline, 2 weeks, 1 month, 2 months, 3 months, 6 months and 12 months. In addition, the rate of change (score) in the ACR50 and DAS28 from the baseline to 2-week, 1-month, 2-month, 6-month, and 12-month follow-up are also the secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Adults with rheumatoid arthritis (score more then 5 of ACR (American College Of Rheumatology) /EULAR (European League Against Rheumatism), 2009 )
* moderate-to-severe disease activity (Disease Activity Score for 28-joint counts (DAS28) of more than 3.2
* an onset of symptoms within 12 months before enrollment, no prior exposure to more than 10mg oral glucocorticoids or biologic agents
* paid employment or unpaid but measurable work (e.g. caring for a family and home)

Exclusion Criteria:

* combined with other disease such as adjuvant arthritis, lupus arthritis, osteoarthritis and et al.
* abnormal liver and my kidney function
* pregnancy or have a plan of pregnancy,breast feeding women
* severe chronic or acute disease interfering with therapy attendance
* alcohol or substance abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of ACR (American College of Rheumatology) 50 | at 3 months
  ACR (American College of Rheumatology) 50 is a standard to describe RA symptoms. ACR 50 is met when the number of tender joints reduces by ≥50%, the number of swollen joints by ≥50%, and at least 3 of the following 5 indexes improves by ≥50%:
  Patient's assessment on arthritis pain using a visual analogue scale (VAS) of 0-100 mm, Patient global assessment on disease activity using VAS scale (0-10), Patient's assessment on physical function and disability (Health Assessment Questionnaire - Disability Index (HAQ-DI)), Acute phase reactant value, such as erythrocyte sedimentation rate (ESR) or C-reactive Protein (CRP) level
changes of The Disease Activity Score (DAS) 28 | from baseline to 3 months
  The DAS28 is an index calculating the number of painful and swollen joints (28 joints, i.e. shoulders, elbows, wrists, metacarpophalangeal and proximal interphalangeal joints, and knees), erythrocyte sedimentation rate and the score of global assessment. The formula of DAS 28 is 0.56×√(28 painful joint count) + 0.28×√(28 swollen joint count) + 0.70× (ln ESR) + 0.014 ×GH. ESR refers to erythrocyte sedimentation rate. GH is the patient's general health visual analog scale (0-10 mm)

SECONDARY OUTCOMES:
changes of The Disease Activity Score (DAS) 28 | from baseline to 2 weeks
  The DAS28 is an index calculating the number of painful and swollen joints (28 joints, i.e. shoulders, elbows, wrists, metacarpophalangeal and proximal interphalangeal joints, and knees), erythrocyte sedimentation rate and the score of global assessment. The formula of DAS 28 is 0.56×√(28 painful joint count) + 0.28×√(28 swollen joint count) + 0.70× (ln ESR) + 0.014 ×GH. ESR refers to erythrocyte sedimentation rate. GH is the patient's general health visual analog scale (0-10 mm)
changes of The Disease Activity Score (DAS) 28 | from baseline to 1 month
  The DAS28 is an index calculating the number of painful and swollen joints (28 joints, i.e. shoulders, elbows, wrists, metacarpophalangeal and proximal interphalangeal joints, and knees), erythrocyte sedimentation rate and the score of global assessment. The formula of DAS 28 is 0.56×√(28 painful joint count) + 0.28×√(28 swollen joint count) + 0.70× (ln ESR) + 0.014 ×GH. ESR refers to erythrocyte sedimentation rate. GH is the patient's general health visual analog scale (0-10 mm)
changes of The Disease Activity Score (DAS) 28 | from baseline to 6 months
  The DAS28 is an index calculating the number of painful and swollen joints (28 joints, i.e. shoulders, elbows, wrists, metacarpophalangeal and proximal interphalangeal joints, and knees), erythrocyte sedimentation rate and the score of global assessment. The formula of DAS 28 is 0.56×√(28 painful joint count) + 0.28×√(28 swollen joint count) + 0.70× (ln ESR) + 0.014 ×GH. ESR refers to erythrocyte sedimentation rate. GH is the patient's general health visual analog scale (0-10 mm)
changes of The Disease Activity Score (DAS) 28 | from baseline to 12 months
  The DAS28 is an index calculating the number of painful and swollen joints (28 joints, i.e. shoulders, elbows, wrists, metacarpophalangeal and proximal interphalangeal joints, and knees), erythrocyte sedimentation rate and the score of global assessment. The formula of DAS 28 is 0.56×√(28 painful joint count) + 0.28×√(28 swollen joint count) + 0.70× (ln ESR) + 0.014 ×GH. ESR refers to erythrocyte sedimentation rate. GH is the patient's general health visual analog scale (0-10 mm)
Rate of ACR (American College of Rheumatology) 50 | at 2 weeks
  ACR (American College of Rheumatology) 50 is a standard to describe RA symptoms. ACR 50 is met when the number of tender joints reduces by ≥50%, the number of swollen joints by ≥50%, and at least 3 of the following 5 indexes improves by ≥50%:
  Patient's assessment on arthritis pain using a visual analogue scale (VAS) of 0-100 mm, Patient global assessment on disease activity using VAS scale (0-10), Patient's assessment on physical function and disability (Health Assessment Questionnaire - Disability Index (HAQ-DI)), Acute phase reactant value, such as erythrocyte sedimentation rate (ESR) or C-reactive Protein (CRP) level
Rate of ACR (American College of Rheumatology) 50 | at 1 month
  ACR (American College of Rheumatology) 50 is a standard to describe RA symptoms. ACR 50 is met when the number of tender joints reduces by ≥50%, the number of swollen joints by ≥50%, and at least 3 of the following 5 indexes improves by ≥50%:
  Patient's assessment on arthritis pain using a visual analogue scale (VAS) of 0-100 mm, Patient global assessment on disease activity using VAS scale (0-10), Patient's assessment on physical function and disability (Health Assessment Questionnaire - Disability Index (HAQ-DI)), Acute phase reactant value, such as erythrocyte sedimentation rate (ESR) or C-reactive Protein (CRP) level
Rate of ACR (American College of Rheumatology) 50 | at 2 months
  ACR (American College of Rheumatology) 50 is a standard to describe RA symptoms. ACR 50 is met when the number of tender joints reduces by ≥50%, the number of swollen joints by ≥50%, and at least 3 of the following 5 indexes improves by ≥50%:
  Patient's assessment on arthritis pain using a visual analogue scale (VAS) of 0-100 mm, Patient global assessment on disease activity using VAS scale (0-10), Patient's assessment on physical function and disability (Health Assessment Questionnaire - Disability Index (HAQ-DI)), Acute phase reactant value, such as erythrocyte sedimentation rate (ESR) or C-reactive Protein (CRP) level
Rate of ACR (American College of Rheumatology) 50 | at 6 months
  ACR (American College of Rheumatology) 50 is a standard to describe RA symptoms. ACR 50 is met when the number of tender joints reduces by ≥50%, the number of swollen joints by ≥50%, and at least 3 of the following 5 indexes improves by ≥50%:
  Patient's assessment on arthritis pain using a visual analogue scale (VAS) of 0-100 mm, Patient global assessment on disease activity using VAS scale (0-10), Patient's assessment on physical function and disability (Health Assessment Questionnaire - Disability Index (HAQ-DI)), Acute phase reactant value, such as erythrocyte sedimentation rate (ESR) or C-reactive Protein (CRP) level
Rate of ACR (American College of Rheumatology) 50 | at 12 months
  ACR (American College of Rheumatology) 50 is a standard to describe RA symptoms. ACR 50 is met when the number of tender joints reduces by ≥50%, the number of swollen joints by ≥50%, and at least 3 of the following 5 indexes improves by ≥50%:
  Patient's assessment on arthritis pain using a visual analogue scale (VAS) of 0-100 mm, Patient global assessment on disease activity using VAS scale (0-10), Patient's assessment on physical function and disability (Health Assessment Questionnaire - Disability Index (HAQ-DI)), Acute phase reactant value, such as erythrocyte sedimentation rate (ESR) or C-reactive Protein (CRP) level
change score of Health Assessment Questionnaire - Disability Index | from baseline to 2 weeks
  The HAQ-DI measure shave eight dimensions of functional activity: pruning, dressing, rising, eating, walking, personal hygiene, reach, grip, and other routine activities. Each item has 4 degrees ranging from 0 to 3. "0" refers to "no functional difficulty", "1" to a bit of functional difficulty, "2" to very much functional difficulty, and "3" to no ability to work. HAQ-DI score 0-1 means mild to moderate functional difficulty; 1-2 means moderate to severe disability; and 2-3 means generally severe disability
change score of Health Assessment Questionnaire - Disability Index | from baseline to 1 month
  The HAQ-DI measure shave eight dimensions of functional activity: pruning, dressing, rising, eating, walking, personal hygiene, reach, grip, and other routine activities. Each item has 4 degrees ranging from 0 to 3. "0" refers to "no functional difficulty", "1" to a bit of functional difficulty, "2" to very much functional difficulty, and "3" to no ability to work. HAQ-DI score 0-1 means mild to moderate functional difficulty; 1-2 means moderate to severe disability; and 2-3 means generally severe disability
change score of Health Assessment Questionnaire - Disability Index | from baseline to 2 months
  The HAQ-DI measure shave eight dimensions of functional activity: pruning, dressing, rising, eating, walking, personal hygiene, reach, grip, and other routine activities. Each item has 4 degrees ranging from 0 to 3. "0" refers to "no functional difficulty", "1" to a bit of functional difficulty, "2" to very much functional difficulty, and "3" to no ability to work. HAQ-DI score 0-1 means mild to moderate functional difficulty; 1-2 means moderate to severe disability; and 2-3 means generally severe disability
change score of Health Assessment Questionnaire - Disability Index | from baseline to 3 months
  The HAQ-DI measure shave eight dimensions of functional activity: pruning, dressing, rising, eating, walking, personal hygiene, reach, grip, and other routine activities. Each item has 4 degrees ranging from 0 to 3. "0" refers to "no functional difficulty", "1" to a bit of functional difficulty, "2" to very much functional difficulty, and "3" to no ability to work. HAQ-DI score 0-1 means mild to moderate functional difficulty; 1-2 means moderate to severe disability; and 2-3 means generally severe disability
change score of Health Assessment Questionnaire - Disability Index | from baseline to 6 months
  The HAQ-DI measure shave eight dimensions of functional activity: pruning, dressing, rising, eating, walking, personal hygiene, reach, grip, and other routine activities. Each item has 4 degrees ranging from 0 to 3. "0" refers to "no functional difficulty", "1" to a bit of functional difficulty, "2" to very much functional difficulty, and "3" to no ability to work. HAQ-DI score 0-1 means mild to moderate functional difficulty; 1-2 means moderate to severe disability; and 2-3 means generally severe disability
change score of Health Assessment Questionnaire - Disability Index | from baseline to 12 months
  The HAQ-DI measure shave eight dimensions of functional activity: pruning, dressing, rising, eating, walking, personal hygiene, reach, grip, and other routine activities. Each item has 4 degrees ranging from 0 to 3. "0" refers to "no functional difficulty", "1" to a bit of functional difficulty, "2" to very much functional difficulty, and "3" to no ability to work. HAQ-DI score 0-1 means mild to moderate functional difficulty; 1-2 means moderate to severe disability; and 2-3 means generally severe disability
change score of Patient Assessment of Arthritis Pain | from baseline to 2 weeks
change score of Patient Assessment of Arthritis Pain | from baseline to 1 month
  VAS score, the range is 0-10, more pain then bigger number
change score of Patient Assessment of Arthritis Pain | from baseline to 2 months
  VAS score, the range is 0-10, more pain then bigger number
change score of Patient Assessment of Arthritis Pain | from baseline to 3 months
  VAS score, the range is 0-10, more pain then bigger number
change score of Patient Assessment of Arthritis Pain | from baseline to 6 months
  VAS score, the range is 0-10, more pain then bigger number
change score of Patient Assessment of Arthritis Pain | from baseline to 12 months
  VAS score, the range is 0-10, more pain then bigger number
change score of Patient Global Assessment of Arthritis | from baseline to 2 weeks
  the range is 0-10, more pain then bigger number
change score of Patient Global Assessment of Arthritis | from baseline to 1 month
  the range is 0-10, more pain then bigger number
change score of Patient Global Assessment of Arthritis | from baseline to 2 months
  the range is 0-10, more pain then bigger number
change score of Patient Global Assessment of Arthritis | from baseline to 3 months
  the range is 0-10, more pain then bigger number
change score of Patient Global Assessment of Arthritis | from baseline to 6 months
  the range is 0-10, more pain then bigger number
change score of Patient Global Assessment of Arthritis | from baseline to 12 months
  the range is 0-10, more pain then bigger number
change score of 36-item Short-Form Health Survey Questionnaire | from baseline to 2 weeks
change score of 36-item Short-Form Health Survey Questionnaire | from baseline to 1 month
  The SF-36 measures eight dimensions, including vitality, body function, body aches, general health perceptions, body functions, emotional function, social function and mental health. SF-36 is widely used in the evaluation of quality of life in patients with rheumatoid arthritis
change score of 36-item Short-Form Health Survey Questionnaire | from baseline to 2 months
  The SF-36 measures eight dimensions, including vitality, body function, body aches, general health perceptions, body functions, emotional function, social function and mental health. SF-36 is widely used in the evaluation of quality of life in patients with rheumatoid arthritis
change score of 36-item Short-Form Health Survey Questionnaire | from baseline to 3 months
  The SF-36 measures eight dimensions, including vitality, body function, body aches, general health perceptions, body functions, emotional function, social function and mental health. SF-36 is widely used in the evaluation of quality of life in patients with rheumatoid arthritis
change score of 36-item Short-Form Health Survey Questionnaire | from baseline to 6 months
  The SF-36 measures eight dimensions, including vitality, body function, body aches, general health perceptions, body functions, emotional function, social function and mental health. SF-36 is widely used in the evaluation of quality of life in patients with rheumatoid arthritis
change score of 36-item Short-Form Health Survey Questionnaire | from baseline to 12 months
  The SF-36 measures eight dimensions, including vitality, body function, body aches, general health perceptions, body functions, emotional function, social function and mental health. SF-36 is widely used in the evaluation of quality of life in patients with rheumatoid arthritis
change score of AIS Sleep Scale | from baseline to 2 weeks
  The Athens Insomnia Scale (AIS) can help patients quantitatively self-evaluate sleep disorders with a psychometric instrument that includes eight indicators for sleep induction, awakenings during the night, final awakening, total sleep duration, sleep quality during the night, wellbeing during the night, functioning capacity during the day time, and sleepiness during the day time. The score for each indicator ranges from 0 to 3, and the total score is 24 points. The higher the score, the worse the sleep quality, and vise versa
change score of AIS Sleep Scale | from baseline to 1 month
  The Athens Insomnia Scale (AIS) can help patients quantitatively self-evaluate sleep disorders with a psychometric instrument that includes eight indicators for sleep induction, awakenings during the night, final awakening, total sleep duration, sleep quality during the night, wellbeing during the night, functioning capacity during the day time, and sleepiness during the day time. The score for each indicator ranges from 0 to 3, and the total score is 24 points. The higher the score, the worse the sleep quality, and vise versa
change score of AIS Sleep Scale | from baseline to 2 months
  The Athens Insomnia Scale (AIS) can help patients quantitatively self-evaluate sleep disorders with a psychometric instrument that includes eight indicators for sleep induction, awakenings during the night, final awakening, total sleep duration, sleep quality during the night, wellbeing during the night, functioning capacity during the day time, and sleepiness during the day time. The score for each indicator ranges from 0 to 3, and the total score is 24 points. The higher the score, the worse the sleep quality, and vise versa
change score of AIS Sleep Scale | from baseline to 3 months
  The Athens Insomnia Scale (AIS) can help patients quantitatively self-evaluate sleep disorders with a psychometric instrument that includes eight indicators for sleep induction, awakenings during the night, final awakening, total sleep duration, sleep quality during the night, wellbeing during the night, functioning capacity during the day time, and sleepiness during the day time. The score for each indicator ranges from 0 to 3, and the total score is 24 points. The higher the score, the worse the sleep quality, and vise versa
change score of AIS Sleep Scale | from baseline to 6 months
  The Athens Insomnia Scale (AIS) can help patients quantitatively self-evaluate sleep disorders with a psychometric instrument that includes eight indicators for sleep induction, awakenings during the night, final awakening, total sleep duration, sleep quality during the night, wellbeing during the night, functioning capacity during the day time, and sleepiness during the day time. The score for each indicator ranges from 0 to 3, and the total score is 24 points. The higher the score, the worse the sleep quality, and vise versa
change score of AIS Sleep Scale | from baseline to 12 months
  The Athens Insomnia Scale (AIS) can help patients quantitatively self-evaluate sleep disorders with a psychometric instrument that includes eight indicators for sleep induction, awakenings during the night, final awakening, total sleep duration, sleep quality during the night, wellbeing during the night, functioning capacity during the day time, and sleepiness during the day time. The score for each indicator ranges from 0 to 3, and the total score is 24 points. The higher the score, the worse the sleep quality, and vise versa
rate of ACR20 | at 2 weeks
rate of ACR20 | at 1 month
  ACR20 is met when ≥20% is achieved in the reduction of tender joint number, swollen joint number, and indexes of 3 of the 5 other measurements
rate of ACR20 | at 2 months
  ACR20 is met when ≥20% is achieved in the reduction of tender joint number, swollen joint number, and indexes of 3 of the 5 other measurements
rate of ACR20 | at 3 months
  ACR20 is met when ≥20% is achieved in the reduction of tender joint number, swollen joint number, and indexes of 3 of the 5 other measurements
rate of ACR20 | at 6 months
  ACR20 is met when ≥20% is achieved in the reduction of tender joint number, swollen joint number, and indexes of 3 of the 5 other measurements
rate of ACR20 | at 12 months
  ACR20 is met when ≥20% is achieved in the reduction of tender joint number, swollen joint number, and indexes of 3 of the 5 other measurements
rate of ACR70 | at 2 weeks
  ACR70 is met when ≥70% is achieved in the reduction of tender joint number, swollen joint number, and indexes of 3 of the 5 other measurements
rate of ACR70 | at 1 month
  ACR70 is met when ≥70% is achieved in the reduction of tender joint number, swollen joint number, and indexes of 3 of the 5 other measurements
rate of ACR70 | at 2 months
  ACR70 is met when ≥70% is achieved in the reduction of tender joint number, swollen joint number, and indexes of 3 of the 5 other measurements
rate of ACR70 | at 3 months
  ACR70 is met when ≥70% is achieved in the reduction of tender joint number, swollen joint number, and indexes of 3 of the 5 other measurements
rate of ACR70 | at 6 months
  ACR70 is met when ≥70% is achieved in the reduction of tender joint number, swollen joint number, and indexes of 3 of the 5 other measurements
rate of ACR70 | at 12 months
  ACR70 is met when ≥70% is achieved in the reduction of tender joint number, swollen joint number, and indexes of 3 of the 5 other measurements

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang Y, Liu Y, Xi Z, Yu Y, Liu L, Mao J, Xiao L, Gu X, Yao M, Cui X, Shi Q, Wang Y, Liang Q. A multicenter, randomized, double-blind, placebo-controlled trial evaluating the efficacy and safety of Huangqi Guizhi Wuwutang granule in patients with rheumatoid arthritis. Medicine (Baltimore). 2019 Mar;98(11):e14888. doi: 10.1097/MD.0000000000014888. PMID 30882703